CLINICAL TRIAL: NCT05950490
Title: Construction of Diagnosis and Treatment System for Primary Vitreoretinal Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Beijing Tongren Hospital (Other); Southern Medical University (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2022-PUMCH-C-038
Record Dates: First submitted 2023-07-11; First posted 2023-07-18 (Actual); Last update posted 2023-07-18 (Actual); Status verified 2023-07

CONDITIONS: Primary Vitreoretinal Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 26 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Cerebrospinal fluid IL-10 was normal
  Interventions: Drug: Intravitreal injection of methotrexate
- Group B: Cerebrospinal fluid IL-10 was normal or elevated
  Interventions: Drug: Intravitreal injection of methotrexate

INTERVENTIONS:
Drug: Intravitreal injection of methotrexate — Intravitreal injection of methotrexate:400ug/0.1mL，Once a week*4 weeks → Once every two weeks*4 weeks → once a month *10 times(16 times a year)
  Systemic therapy:
  Induction period:（Zanubrutinib + Rituximab，ZR） (28 days/cycle) x 6 cycles:Rituximab iv375mg/m2 D1, Zanubrutinib 160mg bid D1-D21; Maintenance treatment:Zanubrutinib 160mg bid x 2 years
  Other Names: Intravitreal injection of methotrexate+systemic therapy

SUMMARY:
This study intends to apply for the establishment of research beds, establish a Chinese PVRL research cohort, and carry out a to achieve the following research objectives:

The goal of this prospective observational study is to construct the diagnosis and treatment system for primary vitreoretinal lymphoma（PVRL）. The study is to achieve the following research objectives:

1. To establish a comprehensive diagnostic criteria for PVRL with high diagnostic efficiency and strengthen the PVRL diagnostic system;
2. To establish a standardized treatment pathway for PVRL and evaluate the efficacy and safety of treatment;
3. To screen the prognosis evaluation indicators, and to establish the follow-up process and prognosis evaluation system of PVRL；
4. To explore the pathogenesis of PVRL, specific tumor markers and drug therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed PVRL patients admitted to the Ophthalmology or Hematology departments of Peking Union Medical College Hospital from 2022 to 2024;
* 18-75 years old;
* The diagnosis was confirmed by pathology, aqueous humor/vitreous IL-10/IL-6, vitreous flow cytometry and gene rearrangement.;
* HIV-Ab negative;
* Creatinine clearance > 50ml/min;
* Sign informed consent.

Exclusion Criteria:

* Combined with other tumors;
* Uncontrolled active infections;
* Pregnant or lactating women;
* Antitumor therapy other than the protocol of this study was used.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed PVRL patients admitted to the Ophthalmology or Hematology departments of Peking Union Medical College Hospital from 2022 to 2024.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Interleukin-10/Interleukin-6（IL-10/IL-6） | 1 year
  aqueous fluid
Interleukin-10/Interleukin-6（IL-10/IL-6） | 2.5 years
  cerebrospinal

CONTACTS AND LOCATIONS:
Overall Officials: Meifen Zhang, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China